CLINICAL TRIAL: NCT00414128
Title: A Randomised Clinical Trial of Mycophenolate Mofetil Versus Cyclophosphamide for Remission Induction in ANCA Associated Vasculitis.
Brief Title: Clinical Trial of Mycophenolate Versus Cyclophosphamide in ANCA Vasculitis
Acronym: MYCYC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Aspreva Pharmaceuticals (Industry); Vifor Pharma (Industry)
Responsible Party: Principal Investigator, David Jayne, Drs David Jayne Consultant in Nephrology and Vasculitis, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MYCYC; Eudract: 2006-001663-33
Record Dates: First submitted 2006-12-19; First posted 2006-12-21 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Vasculitis
Keywords: vasculitis; ANCA; mycophenolate mofetil; cyclophosphamide; Anti neutrophil cytoplasm antibody associated vasculitis
MeSH Terms: conditions — Vasculitis | interventions — Mycophenolic Acid; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mycophenolate mofetil (Experimental): Mycophenolate mofetil for 3-6 months until in stable remission, dose 2-3g/day
  Interventions: Drug: mycophenolate mofetil
- cyclophosphamide (Active Comparator): pulsed intravenous cyclophosphamide 15mg/kg for 3-6 months (6-10 doses)until in stable remission
  Interventions: Drug: cyclophosphamide

INTERVENTIONS:
Drug: mycophenolate mofetil — 2-3g/day for 3-6 months, in tablet, capsule or liquid form
  Other Names: Cellcept
  Arms: mycophenolate mofetil
Drug: cyclophosphamide — intravenous cyclophosphamide, 15mg/kg with dose reductions according to age and renal function, for 3-6 months (6-10 doses total)
  Other Names: cytoxan
  Arms: cyclophosphamide

SUMMARY:
The purpose of this study is to investigate whether mycophenolate mofetil is effective as treatment for new cases of ANCA associated vasculitis.

DETAILED DESCRIPTION:
There is a clear need for improved therapy in ANCA associated vasculitis where current treatments are toxic and contribute to poor outcomes. Conventional therapy combines cyclophosphamide with prednisolone but is associated with severe adverse events in 35%, early mortality, malignancy and infertility. Mycophenolate mofetil (MMF) is a newer immunosuppressive drug which has superior efficacy to azathioprine in solid organ transplantation. MMF is an effective alternative to cyclophosphamide in lupus nephritis. Open label studies and retrospective surveys point to the efficacy and low toxicity of MMF in vasculitis.

We hypothesise that MMF not be less effective than cyclophosphamide for remission induction in AASV. 140 new patients will be randomised to MMF 3g/day or a European consensus intravenous cyclophosphamide regimen, with the same prednisolone dosing. Following a six month induction course all patients will receive consensus remission maintenance treatment with azathioprine and prednisolone. The primary end-point will be remission rate by six months, secondary end-points include relapse rate at 18 months and safety. The trial will be conducted in 10 countries by members of the European Vasculitis Study Group (EUVAS). The trial duration will be 42 months (24 months recruitment, 18 months follow up).

ELIGIBILITY:
Inclusion Criteria:

Inclusion (requires all):

* New diagnosis of AASV (WG or MPA) (within the previous six months)
* Active disease (defined by at least one major or three minor BVAS 2003 items, see appendix 1)
* ANCA positivity (c-ANCA and PR3-ANCA or p-ANCA and MPO-ANCA) or histology confirming active vasculitis from any organ (see appendix )
* Written informed consent

Exclusion Criteria:

* Previous treatment with:

  * MMF: more than two weeks ever.
  * Cyclophosphamide: more than two weeks daily oral or more than 1 pulse of IV CYC (15mg/kg)
  * Rituximab or high dose intravenous immunoglobulin within the last twelve months
* Active infection (including hepatitis B, C, HIV and tuberculosis).
* Known hypersensitivity to MMF, AZA or CYC.
* Cancer or an individual history of cancer (other than resected basal cell skin carcinoma).
* Females who are pregnant, breast feeding, or at risk of pregnancy and not using a medically acceptable form of contraception.
* Any condition judged by the investigator that would cause the study to be detrimental to the patient.
* Any other multi-system autoimmune disease including Churg Strauss angiitis, SLE, anti GBM disease and cryoglobulinaemia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2007-03; Primary Completion 2011-07 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Remission rates at 6 months | 6 months
  Assessed by BVAS score of zero on 2 consecutive assessments

CONTACTS AND LOCATIONS:
Overall Officials: David Jayne, Principal Investigator — Addenbrooke's Hospital, Cambridge, UK; Lorraine Harper, Principal Investigator — Birmingham University, UK; Rachel Jones, Principal Investigator — Addenbrooke's Hospital, UK
Locations (1):
- Addenbrookes Hospital, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Derived] Jones RB, Hiemstra TF, Ballarin J, Blockmans DE, Brogan P, Bruchfeld A, Cid MC, Dahlsveen K, de Zoysa J, Espigol-Frigole G, Lanyon P, Peh CA, Tesar V, Vaglio A, Walsh M, Walsh D, Walters G, Harper L, Jayne D; European Vasculitis Study Group (EUVAS). Mycophenolate mofetil versus cyclophosphamide for remission induction in ANCA-associated vasculitis: a randomised, non-inferiority trial. Ann Rheum Dis. 2019 Mar;78(3):399-405. doi: 10.1136/annrheumdis-2018-214245. Epub 2019 Jan 5. PMID 30612116
- See also: EUVAS web site — http://vasculitis.org